CLINICAL TRIAL: NCT03269851
Title: Radiological Parameters Predicting Neurological Injury After Thoracolumbar Spinal Fractures
Brief Title: Parameters of Neurological Deficit After Thoracolumbar Fractures
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zamboo Safwat, Principal investigator, Assiut University
Other Study IDs: Neurological deficit; Thoracolumbar fractures (Other: Assiut University Hospital)
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: SPINAL Fracture
Keywords: neurological deficit
MeSH Terms: conditions — Spinal Fractures; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: computed tomography — ct will be done to detect radiological risk factors for neurological deficits after thoracolumbar fractures

SUMMARY:
To detect Radiological parameters affecting neurological injury after thoracolumbar spinal fractures.

DETAILED DESCRIPTION:
Thoracolumbar spine fractures are the most common spinal column fractures. High activity and lack of stability make it more prone to fractures.

Many studies have attempted to determine whether the neurological deficit in such fractures is related to spinal canal stenosis or other parameters observed on axial computed tomography (CT). However, this relationship remains controversial.

Few reports shed light on the relation between different imaging parameters like sagittal alignment, vertebral body compression, canal stenosis, and type of fracture according to AO classification with the severity of nerve damage.

These four radiographic parameters will be tested as expected risk factors for the neurological deficit in thoracolumbar fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with Acute (within one month) thoracolumbar spine fracture above 18 years old with or without neurological deficit
2. In orthopaedics and trauma department of Assiut university hospital from 1st of November 2018 to 31 st of October 2019.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients suffering from preoperative neurological diseases that hinder our examination like peripheral neuropathy or previous strokes.
* Obtuned patients who cannot be properly examined like those with low GCS score.
* Patients with old thoracolumbar fractures more than one month duration.
* Patients with pathological spine fractures like those with osteoporosis and cancer metastasis.
* Patients with fracture type A0 according to AO classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with Acute (within one month) thoracolumbar spine fracture above 18 years old with or without neurological deficit in orthopaedics and trauma department of Assiut university hospital from 1st of November 2018 to 31 st of October 2019.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
To Measure spinal canal stenosis by cubic cm | one year
  CT-Radiological parameters measured in patients with or without thoracolumbar fractures .
To measure sagittal alignment of vertebral column by cobb angle | one year
  CT-Radiological parameters measured in patients with or without thoracolumbar fractures
To measure vertebral body compression by cm | one year
  CT-Radiological parameters measured in patients with or without thoracolumbar fractures
To measure type of fracture according to AO classification | one year
  CT-Radiological parameters measured in patients with or without thoracolumbar fractures

SECONDARY OUTCOMES:
Proportion of Neurological deficit among patients with thoracolumbar spine fractures. | one year
  Number of patients with neurological deficit to the total number of patients with thoracolumbar spine fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed G. Hassan, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- See also: The significance of thoracolumbar spinal canal size in spinal cord injury patients. — https://doi.org/10.1097/00007632-200102150-00013
- See also: CT scan prediction of neurological deficit in thoracolumbar burst fractures. — http://bjj.boneandjoint.org.uk/content/74-B/5/683.short
- See also: Relationship between traumatic spinal canal stenosis and neurologic deficits in thoracolumbar burst fractures. — https://doi.org/10.1097/00007632-198811000-00011
- See also: Neurologic injury and recovery in patients with burst fracture of the thoracolumbar spine. — https://doi.org/10.1097/00007632-199902010-00020
- See also: Correlation among canal compromise, neurologic deficit, and injury severity in thoracolumbar burst fractures. — https://doi.org/10.1097/01.brs.0000231730.34754.9e